CLINICAL TRIAL: NCT03384147
Title: Metabolic Imprints of Alcoholic Beverages
Acronym: MetAl
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Carlsberg Foundation (Unknown)
Responsible Party: Principal Investigator, Professor Lars Ove Dragsted, Professor, Head of Section, University of Copenhagen
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: M228
Record Dates: First submitted 2017-12-11; First posted 2017-12-27 (Actual); Last update posted 2017-12-27 (Actual); Status verified 2017-12

CONDITIONS: Metabolic Side Effects of Drugs and Substances
MeSH Terms: conditions — Metabolic Side Effects of Drugs and Substances | interventions — Drinking

STUDY DESIGN:
Intervention Model Description: The study was conducted in two predefined groups of volunteers, 1) daily alcohol users of maximally one (females) or two (males) drinks per day, and 2) occasional drinkers (0-2 drinks per week). Group 1 was asked to abstain from alcohol for 3 weeks, then to resume drinking 1-2 drinks daily for the next three weeks. Group 2 was asked to drink 1-2 drinks daily for 3 weeks and then to abstain for the following 3 weeks. During the alcohol intake period both groups were randomized to sequences of 4-5 days with red wine, white wine, lager beer, apple cider, or spirits. The primary endpoint was an effect of alcohol on dihydroepiandrosterone sulphate excretion in urine. Biomarkers of alcohol intake and alcohol-induced metabolic change, physical activity, or well-being were secondary outcomes.
Masking Description: Intake of alcoholic drinks or abstaining cannot be masked to participants or care providers (delivering the alcoholic beverages). The outcomes included biomarkers of alcohol intake so in practice the investigator and outcomes assessor could not be blinded either.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drinking (Experimental): Occasional drinkers assigned to start with a 3week drinking period (women 1 u/day - men 2 u/day)
  Followed by crossover without washout to 3 week abstaining period
  Interventions: Dietary Supplement: Drinking; Other: Abstaining
- Abstaining (Experimental): Habitual drinkers assigned to start 2 weeks of abstaining from alcohol
  Followed by crossover without washout to 3 weeks drinking (women 1 u/day - men 2 u/day)
  Interventions: Dietary Supplement: Drinking; Other: Abstaining

INTERVENTIONS:
Dietary Supplement: Drinking — Five different types of alcohol given to participants for 4-5 days in a random sequence for 3 weeks
Other: Abstaining — Participants are abstaining from all alcoholic beverages for three weeks

SUMMARY:
Metabolic imprints of five different types of alcohol will be investigated in two study groups.

The study will be an assessor-blinded, parallel dietary trial (crossover design).

The project aims to identify the chemical nature and kinetics of metabolite changes related to alcohol, hops, grapes and other beverage constituents as well as the brewing processes.

DETAILED DESCRIPTION:
Metabolic imprints of five different types of alcohol will be investigated in two study groups of 15 participants in each with equal distribution of gender, occasional (0-2 u/week) and habitual drinkers (>2 u/week), respectively.

The intervention is divided into two periods: abstaining and drinking period. Occasional drinkers begin the abstaining intervention and habitual drinkers begin the drinking intervention, and cross-over after 3 weeks.

In the drinking period women consume 1 unit/day and men 2 units/day.

Study participants will consume five different types of alcohol; beer, cider, white wine, red wine and spirits. The sequence of alcohol consumption in the drinking period is randomized by 'random number allocation'.

Study participants are asked to collect 24h urine samples three days in beginning of each intervention and one day in the end of last intervention. The remaining days of the trial they are asked to make a urine spot test each morning at home. Beside urine samples, they are to give blood samples on each trial day and at screening (6 times). Overnight-fasting blood samples are drawn at day 0, 1 and 21, 22 and 42 of the six week intervention and one at screening before intervention.

Furthermore, participants receive kits to provide a dry blood sampling the following three days after trial days in situ. There will also be taken blood pressure and questionnaire handouts. A voluntary hair sample will be taken at Baseline (day 0) and final day of intervention (day 42).

From these samples the following will be determined:

1. dehydroepiandrosterone sulphate (DHEAS) and related (steroid) hormones and metabolites (primary hypothesis is a sustained increase in DHEAS following alcohol intake)
2. cresol, cresol sulphate, indoxyl sulphate and indole acetic acid (human microbial co-metabolites)
3. humulone-derived conjugates and several analogues and unidentified metabolites from the intake of raw materials from beverage production, including hops, malt, cider apples and grapes etc. (by explorative methods)
4. malt- or brewing-related unidentified metabolites (by explorative methods)
5. additional markers of wine and strong liquor intake (by explorative methods)
6. investigating the use of sampling urine and blood on filter papers and the feasibility of collecting small hair samples
7. investigating metabolic markers in relation to blood pressure, heart rate, physical activity, blood lipids, fibrinogen, adiponectin, and psychosocial well-being etc. after 3 weeks light to moderate alcohol intake or abstaining.
8. metabolic profiling of urine, blood and hair to explore contrasts between periods of drinking and abstaining or periods with specific alcoholic beverages.

ELIGIBILITY:
Inclusion Criteria:

* 20 years of age
* No intolerance of alcohol
* Experience with alcohol
* Able to use smartphone or tablet

Exclusion Criteria:

* Serious chronic health conditions or psychiatric diseases
* Chronic intake of medicine (beside birth control and SSRI)
* Alcohol and/or drug abuse assessed AUDIT score >4 (AUDIT = Alcohol Use Disorders Identification Test).
* Blood samples/donations during trial and 3 months prior
* Liver dysfunction
* High risk of breast cancer assessed by BCRAT score (BCRAT = The Breast Cancer Risk Assessment Tool)
* Pregnancy or lactating

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-01-13 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
DHEAS | 3 weeks
  Changes in dehydroepiandrosterone sulphate (DHEAS) and related (steroid) hormones and metabolites

SECONDARY OUTCOMES:
Markers of alcohol intake | 3 weeks
  Ethyl glucuronide, ethyl sulphate, fatty acid ethyl esters, phosphatidyl ethanol and any other ethanol metabolite
Human microbial co-metabolites | 3 weeks
  Cresol, cresol sulphate, indoxyl sulphate and indole acetic acid
Markers of intake of raw materials from the beverage productions | 1 day
  Humulone-derived conjugates and several analogues and unidentified metabolites from the intake of raw materials used in beverage production, including hops, malt, cider apples, grapes, unknown metabolites from processing, etc.
Metabolites from outcomes 1-4 measured in dry urine spots | 1 day
  Investigating the use of sampling urine on cotton sticks
Metabolites from outcomes 1-4 measured in dry blood samples | 1 day
  Investigating the use of sampling blood on filter papers
Metabolites from outcomes 1-4 measured in a hair sample | 3 weeks (1 day)
  Investigating the feasibility of collecting small hair samples before and after trial
Blood pressure | 1d - 3 weeks
  Investigating changes in blood pressure and heart rate from beginning to end of each intervention period.
Physical activity monitoring | 1d - 3weeks
  Investigating changes in physical activity from beginning to end of each intervention period using a chip with a 3D-gyro mounted on the thigh to record movements during periods of 24-72 hours at the beginning and end of the intervention periods.
Blood lipids | 3 weeks
  Investigating changes in blood lipids at the end of each intervention period
Fibrinogen | 3 weeks
  Investigating changes in fibrinogen and related coagulation factors at the end of each intervention period
Adiponectin | 3 weeks
  Investigating changes in adiponectin at the end of each intervention period
Psychosocial well-being | 3 weeks
  Investigating changes in psycho-social well-being using a standardized questionnaire at the beginning and end of each intervention period.

OTHER OUTCOMES:
Discriminant metabolic profiles | 3 weeks
  Metabolic profiles of blood, urine or hair discriminating periods of alcohol drinking and abstaining determined by receiver-operator characteristics of prediction models provided by partial least squares discriminant analyses comparing random training and test sets.
Discriminant metabolic profiles | 4-5 days
  Metabolic profiles of dry urine spots discriminating periods of drinking specific alcoholic beverages (beer, cider, red wine, white wine or spirits) with abstaining determined by receiver-operator characteristics of prediction models provided by partial least squares discriminant analyses comparing random training and test sets.

CONTACTS AND LOCATIONS:
Overall Officials: Lars O Dragsted, PhD, Principal Investigator — University of Copenhagen
Locations (1):
- Department of Nutrition, Exercise and Sports, University of Copenhagen, Copenhagen, Frederiksberg C, Denmark

IPD SHARING:
Plan to Share IPD: Yes
After study completion the participant ID's will be anonymized to allow data sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 3-6 months after publication of data in a peer reviewed journal when the study has been fully anonymized.
Access Criteria: Through the web-site, https://enpadasi.science.ku.dk/

REFERENCES:
- [Derived] Wilkens TL, Ziegler Z, Aru V, Khakimov B, Overgaard SL, Engelsen SB, Dragsted LO. 1-2 Drinks Per Day Affect Lipoprotein Composition after 3 Weeks-Results from a Cross-Over Pilot Intervention Trial in Healthy Adults Using Nuclear Magnetic Resonance-Measured Lipoproteins and Apolipoproteins. Nutrients. 2022 Nov 27;14(23):5043. doi: 10.3390/nu14235043. PMID 36501072